CLINICAL TRIAL: NCT06548919
Title: Effectiveness and Safety of Different Treatment Regimens in Patients With ESR1-mutated HR+/HER2-advanced Breast Cancer After Failure of Prior Endocrine Therapy: a Prospective, Non-interventional, Real-world Study
Brief Title: Current Status of Treatment for Chinese Patients With ESR1-mutated HR+/HER2-advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ABC-RWS-02
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: ESR1 Gene Mutation; Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy
  Interventions: Drug: Endocrine therapy
- Endocrine therapy
  Interventions: Drug: Chemotherapy Prednisone

INTERVENTIONS:
Drug: Endocrine therapy — All endocrine treatment regimens approved for advanced breast cancer, including tamoxifen, aromatase inhibitors, fulvestrant, etc.
  Groups: Chemotherapy
Drug: Chemotherapy Prednisone — All chemotherapy treatment regimens approved for advanced breast cancer
  Groups: Endocrine therapy

SUMMARY:
This is a prospective, non-interventional real-world study to observe the efficacy and safety of different treatment regimens in patients with ESR1-mutated HR+/HER2-advanced breast cancer after failure of endocrine therapy.

Epidemiological data, efficacy and safety measures will be collected for each subject. Data on efficacy and safety assessment indicators will be collected every 2-3 months until disease progression, receipt of a new anti-tumour treatment modality, death, loss to follow-up, and arrival at the data collection cut-off date. The cut-off date for data collection is defined as 8 weeks after completion of 6 visits for each subject, or 4 weeks after treatment discontinuation and subject discontinuation/withdrawal. Subjects receiving a different treatment regimen remained subject to assessment of safety indicators 4 weeks after discontinuation of the original treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* 1. must have a histologically or cytologically confirmed diagnosis of breast cancer with evidence of locally advanced disease unsuitable for excision or radical radiotherapy, or evidence of metastatic disease unsuitable for radical treatment.
* 2. female ≥ 18 years of age
* 3. female subjects must be postmenopausal (meeting any of the following criteria is sufficient) a) Has undergone oophorectomy. b) Age ≥ 60 years. c) 40 years old < age ≤ 60 years old with 1 year of menopause. d) Age <60 years and receiving ovarian suppression therapy.
* 4. ER-positive and HER2-negative status and ESR1-mutation positive must be confirmed.
* 5. must have progressed on at least one line of endocrine therapy prior to enrollment, including monotherapy or combination therapy.
* 6. have normal organ function (as assessed by the investigator).

Exclusion Criteria:

* 1. women who are pregnant or breastfeeding
* 2. known difficulties in tolerating oral medications, or conditions that interfere with the absorption of oral medications or allergies to medications and their excitements
* 3. other conditions that make enrollment in the study unsuitable, at the discretion of the investigator

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with HR+/HER2-advanced breast cancer with ESR1 mutation after failure of endocrine therapy
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 18 months
  Progression-free survival

SECONDARY OUTCOMES:
ORR | 6 months
  Objective response rate
CBR | 6 months
  Clinical benefit rate
DoR | 18 months
  Duration of response

OTHER OUTCOMES:
Adverse event rate | 18 months
  Percentage of occurrences of adverse events
Serious adverse event rate | 18 months
  Percentage of occurrences of serious adverse events
Treatment regimen | 18 months
  Proportion of endocrine therapy, endocrine-targeted combination therapy or chemotherapy
Medication adherence | 18 months
  proportion of days covered

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Haidafu Internet Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No